CLINICAL TRIAL: NCT03443154
Title: Vaginal Fluid (VF) Test VF-Test™ for Prediction of Extremely Preterm Birth After Exam-Indicated Cerclage Protocol for Prospective, Multicenter, Cohort Clinical Trial
Brief Title: VF Test for Prediction of Extremely PTB After Cerclage
Status: Withdrawn | Type: Observational
Why Stopped: Industry sponsor withdrew financial support as well as the testing equipment.
Sponsor: Pediatrix (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OBX0039
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-02

CONDITIONS: Preterm Birth; Infection
Keywords: Cerclage; Preterm birth
MeSH Terms: conditions — Premature Birth; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: VF-Test — A vaginal fluid test of interleukin-6 (IL-6) and alphafetoprotein (AFP).
  Other Names: vaginal fluid test.

SUMMARY:
The purpose of this research study is to determine if a vaginal fluid (VF) test can predict very early preterm birth in patients who are scheduled to have an exam indicated cerclage for severe cervical shortening.

Prior to participants undergoing a scheduled amniocentesis two swabs to collect vaginal secretions for the VF tests will be done. During the amniocentesis your doctor will remove amniotic fluid as part of the routine clinical care. From that fluid sample, the study will use less than a quarter teaspoon for the amniotic fluid study test (AF test). Data regarding maternal and birth outcomes will be collected by medical record review.

DETAILED DESCRIPTION:
The purpose of this research study is to determine if a vaginal fluid (VF) test can predict very early preterm birth in patients who are scheduled to have an exam indicated cerclage for severe cervical shortening.

Prior to participants undergoing a scheduled amniocentesis, an ultrasound will be done to confirm cervical length and dilation. During a separate sterile speculum exam, the physician will use two swabs to collect vaginal secretions for the VF test. During the amniocentesis the doctor will remove approximately 2 teaspoon of amniotic fluid as part of your standard clinical care. From that fluid sample, the study will use less than a quarter teaspoon for a amniotic fluid study test (AF test). Data regarding maternal and birth outcomes will be collected by medical record review.

The vaginal fluid (VF) sample collection will take approximately 15 minutes to do. The total time in the study is about seven and a half months (from the time the patient consents until 4 weeks after delivery). The only study procedure the patient will experience during her study participation is the collection of the vaginal fluid specimens.

ELIGIBILITY:
Inclusion Criteria:

* Participant age 18 years or older
* Gestational age between 16w0d to 25w6d
* Singleton fetus with no apparent major anomalies on ultrasound exam
* Sonographically absent cervical length and/or sterile digital exam of 2cm or greater dilation
* Exam-indicated cervical cerclage has been recommended by clinician and patient agrees to proceed with cervical cerclage placement
* Decision has been made by provider to perform pre-cerclage amniocentesis to rule-out infection, with the understanding that cerclage is contraindicated if findings indicate probable or definitive infection, and patient agrees.

Exclusion Criteria:

* Planned termination of pregnancy
* Clinical features consistent with placental abruption or chorioamnionitis
* Need for immediate delivery based on maternal or fetal issues
* Fetus with ultrasound-determined major congenital anomalies
* Multiple gestation
* Rupture of membranes
* Patient does not give consent to participate in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital based patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of very preterm birth (PTB) | Time frame measured on the date of infant was born. We anticipate this time frame to be approximately 20 weeks.
  Rate of Very PTB (PTB at less than 28 weeks of pregnancy)

SECONDARY OUTCOMES:
Rate of Delivery within 7 days of cervical cerclage | Time frame measured from the date the cerclage was placed until 7 days later
  Rate of Delivery within 7 days of cervical cerclage placement
Rate of Delivery at later than 34 weeks of pregnancy | Time frame measured from the time the patient reaches 34 weeks 1 day of pregnancy until birth
  Rate of Delivery at later than 34 weeks of pregnancy (ie. 34 week pregnant until 42 weeks)
Rate of a positive VF test results in association with adverse maternal and perinatal outcomes. | Time frame measured from the time of VF test until 28 days after delivery.
  Rate of a positive VF test results in association with adverse maternal and perinatal outcomes. (defined as death or one or more pre-specified morbidities)
Comparison of AF Test and VF Test results in prediction of a positive amniotic fluid culture | Time frame measured at the time of the amniocentesis
  Comparison of amniotic fluid (AF) Test and vaginal fluid (VF) Test results in prediction of a positive amniotic fluid culture

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Vanderhoeven, MD, Principal Investigator — Pediatrix

IPD SHARING:
Plan to Share IPD: Undecided
Not decided at this time